CLINICAL TRIAL: NCT03810092
Title: Analysis of the Relationship Between Early Postoperative Anemia and the Evolution of Autonomy at 6 Months in Patients 75 Years of Age and Older Operated on Following a Fracture of the Upper End of the Femur
Acronym: PAAF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD117-17
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Femoral Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fracture of the upper extremity of the femur is a condition whose frequency increases with age. It is a serious disease, with multiple consequences such as a decrease in life expectancy, quality of life and patient autonomy. In this observational study, the investigators wish to evaluate the evolution of the autonomy of very elderly patients operated on for an upper extremity femur fracture as a function of early post-operative anemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Patient operated on a fracture of the upper extremity of the femur
* Patient, family or close relative who does not object to participation in the study
* Patient affiliated to a social security system
* Patient who can be monitored as part of the protocol

Exclusion Criteria:

* Refusal to participate in the study (patient, family or trusted relative)
* Patient with support on the operated limb not authorized by the surgeon
* Patient with an associated fracture (polytrauma, concomitant trauma to the upper limb...)
* Patient with a pathologic fracture
* Patient included in Category 1 interventional research (involving a drug or medical device)
* Patient deprived of liberty
* Patient not affiliated to a social security system

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study is intended for patients over 75 years of age who have had a fracture of the upper extremity of the femur operated on.
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Romain DECOURS, Principal Investigator — CHD Vendée
Locations (5):
- France (5):
  - CHU Angers, Angers
  - CH Cholet, Cholet
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH Saint Malo, St-Malo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent to Treat Population: Patients 75 Years of Age and Older Operated on Following a Fracture of the Upper End of the Femur
Period: Overall Study
Arm/Group | Intent to Treat Population
Started | 255
Completed | 195
Not Completed | 60
Not completed — no ground support | 17
Not completed — ADL not done at J0 | 16
Not completed — No hemoglobin measure at J5 | 27

BASELINE CHARACTERISTICS:
Arm/Group | Intent to Treat Population
Number analyzed (Participants) | 238
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 88 [83 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181
  Male | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Median (Inter-Quartile Range); unit: kg/m²] — Population: Missing value
  kg/m²
    number analyzed (Participants) | 235
    (all) | 23 [20.9 to 25.7]
Anterior fracture [Count of Participants; unit: Participants] | 81
Hospitalisation time [Median (Inter-Quartile Range); unit: days] | 6 [5 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Rate
Time Frame: 5 days after surgery
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Intent to Treat Population
Number analyzed (Participants) | 159
g/dl | 10 [9.2 to 10.9]

2. Primary Outcome: Questionnaire Activities of Daily Living
Description: For each question, a point from 0 (worst value) to 1 (best value) is assigned. The total score is 6 points.
  A loss of autonomy will be defined by the decrease of one or more points in the ADL.
  Result showed here is the difference of ADL score intra patient
Time Frame: Pre-fractural and 6 months after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intent to Treat Population
Number analyzed (Participants) | 181
score on a scale | 1 [0.5 to 2]
Statistical Analysis 1: Comparison: Intent to Treat Population; Relationship between ADL score evolution and hemoglobine rate, in the no transfusion group; Test type: Other; p = 0.05, Regression, Linear; Odds Ratio, log = -0.04, 95% CI 2-sided [-0.55 to 0.42]
Statistical Analysis 2: Comparison: Intent to Treat Population; Relationship between ADL score evolution and hemoglobine rate, in the transfusion group; Test type: Other; p = 0.05, Regression, Logistic; Odds Ratio, log = 0.39, 95% CI 2-sided [-1 to 2.2]

ADVERSE EVENTS:
Time Frame: Time lenght is between inclusion and 6 month after baseline
Arm/Group | Intent to Treat Population
All-Cause Mortality (participants affected / at risk) | 37/238
Serious Adverse Events (participants affected / at risk) | 0/238
Other Adverse Events (participants affected / at risk) | 0/238

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT03810092/Prot_SAP_000.pdf